CLINICAL TRIAL: NCT00263926
Title: Immunotherapy of Wasp Venom Allergy: Comparison of a Purified Preparation to Conventional Aqueous Wasp Venom in an Open Controlled Study
Brief Title: Efficacy and Safety of a Purified Standardised Wasp Venom Preparation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergopharma GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Al1000ig
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Allergy
Keywords: Wasp venom allergy,; specific immunotherapy
MeSH Terms: conditions — Hypersensitivity; Venom Hypersensitivity | interventions — Wasp Venoms

INTERVENTIONS:
Biological: wasp venom

SUMMARY:
The trial is performed to assess efficacy and safety of a purified standardised wasp venom preparation in wasp venom allergy

ELIGIBILITY:
Inclusion Criteria:

* History of wasp venom allergy,
* Positive RAST to wasp venom,
* Positive skin prick test to wasp venom

Exclusion Criteria:

* Serious chronic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-03; Primary Completion 2007-05 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annemie Narkus, M.D., Principal Investigator
Locations (1):
- Allergopharma GmbH & Co. KG, Reinbek, Germany

REFERENCES:
- See also: Leader in specific allergy research and therapy — http://www.allergopharma.de